CLINICAL TRIAL: NCT00371319
Title: To Compare the Efficacy of Tacrolimus and Mycophenolate Mofetil for the Initial Therapy of Active Lupus Nephritis
Brief Title: Comparing the Efficacy of Tacrolimus and Mycophenolate Mofetil for the Initial Therapy of Active Lupus Nephritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tuen Mun Hospital (Other Government)
Responsible Party: Principal Investigator, Chi Chiu Mok, Consultant, Tuen Mun Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HARECCTR0500018
Record Dates: First submitted 2006-09-01; First posted 2006-09-04 (Estimated); Last update posted 2014-07-02 (Estimated); Status verified 2014-07

CONDITIONS: Lupus Nephritis
Keywords: lupus; nephritis; tacrolimus; mycophenolate mofetil
MeSH Terms: conditions — Lupus Nephritis; Nephritis | interventions — Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tacrolimus (Active Comparator): Tacrolimus treatment
  Interventions: Drug: tacrolimus
- mycophenolate mofetil (Active Comparator): mycophenolate mofetil
  Interventions: Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: tacrolimus — 0.06-0.1 mg/kg/day
  Other Names: Prograf
  Arms: Tacrolimus
Drug: mycophenolate mofetil — 2-3 gm/day
  Other Names: Cellcept
  Arms: mycophenolate mofetil

SUMMARY:
The purpose of this study is comparing the efficacy of tacrolimus and mycophenolate mofetil for the initial therapy of active lupus glomerulonephritis.

DETAILED DESCRIPTION:
Patients with biopsy proven active lupus nephritis will be randomized to receive tacrolimus or mycophenolate mofetil, on top of corticosteroids, for initial treatment. Efficacy and adverse effects will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who fulfill at least 4 of the ACR criteria for SLE
2. Age >= 18 years
3. Biopsy proven active lupus glomerulonephritis (ISN/RPS class III/IV/V)
4. Serum creatinine < 200 umol/L at the time of randomization

Exclusion Criteria:

1. Patients who refuse to be randomized for treatment
2. Patients who prefer treatment with conventional agents such as oral or intravenous CYC for various reasons
3. Serum creatinine >= 200 umol/L at the time of randomization
4. Patients without renal biopsy or those who have lupus nephritis ISN/RPS class I,II,VI
5. Patients who are pregnant or plan for pregnancy within 12 months after randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2005-09; Primary Completion 2014-05 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
remission rate | month 6

SECONDARY OUTCOMES:
renal function deterioration, relapse and mortality | month 60

CONTACTS AND LOCATIONS:
Overall Officials: CC MOK, MD, FRCP, Principal Investigator — Tuen Mun Hospital Hong Kong
Locations (1):
- Tuen Mun Hospital, Hong Kong, China

REFERENCES:
- [Derived] Mok CC, Ho LY, Ying SKY, Leung MC, To CH, Ng WL. Long-term outcome of a randomised controlled trial comparing tacrolimus with mycophenolate mofetil as induction therapy for active lupus nephritis. Ann Rheum Dis. 2020 Aug;79(8):1070-1076. doi: 10.1136/annrheumdis-2020-217178. Epub 2020 May 24. PMID 32448782
- [Derived] Mok CC, Ying KY, Yim CW, Siu YP, Tong KH, To CH, Ng WL. Tacrolimus versus mycophenolate mofetil for induction therapy of lupus nephritis: a randomised controlled trial and long-term follow-up. Ann Rheum Dis. 2016 Jan;75(1):30-6. doi: 10.1136/annrheumdis-2014-206456. Epub 2014 Dec 30. PMID 25550339